CLINICAL TRIAL: NCT00357032
Title: A Phase 2 Study of PXD101 in Patients With Relapsed or Refractory Acute Myelogenous Leukemia or Patients Over 60 With Newly-Diagnosed Acute Myelogenous Leukemia
Brief Title: PXD101 in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02838; PHII-68; N01CM62209 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — belinostat

ARMS (1):
- Treatment (belinostat) (Experimental): Patients receive PXD101 IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 6-12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: belinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well PXD101 works in treating patients with relapsed or refractory acute myeloid leukemia or older patients with newly diagnosed acute myeloid leukemia. PXD101 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the response rate (complete response and partial response) in patients with acute myeloid leukemia treated with PXD101.

SECONDARY OBJECTIVES:

I. Evaluate the overall survival of these patients. II. Evaluate the duration of response in these patients. III. Evaluate the toxicity of this drug in these patients.

TERTIARY OBJECTIVES:

I. Evaluate molecular response to PXD101.

OUTLINE:

Patients receive PXD101 IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 6-12 months in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples are obtained before and after study treatment for laboratory studies.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed acute myelogenous leukemia
* The diagnosis must be made by bone marrow aspirate and biopsy; patients must have routine cytochemical evaluation along with immunophenotyping done by flow cytometry; cytogenetic analysis must also be performed
* For patients age 18-59 years, at least one prior regimen of induction chemotherapy is required; patients who have been treated with bone marrow or stem cell transplantation are eligible; there is no prior therapy requirement for patients age > 60

  * Patients for whom potentially curative treatment is available must be offered this treatment and decline
* Life expectancy of greater than 3 months
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Serum total bilirubin =< 2.0 mg/dl
* AST and ALT =< 2.5 times upper limit of normal (ULN)
* Creatinine clearance >= 60 mL/min OR creatinine < 1.5 times ULN
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of PXD101 will be determined following review of their case by the principal investigator

  * Efforts should be made to switch patients with gliomas or brain metastases who are taking enzyme inducing anticonvulsant agents to other medications
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients taking hydroxyurea for the purpose of cytoreduction should discontinue this medication at least 24 hours prior to the initiation of therapy with PXD101

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known central nervous system (CNS) disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101
* Patients may not have had prior treatment with another HDAC inhibitor within 1 week of initiation of therapy with PXD101; patients receiving valproic acid should stop this medication at least 1 week prior to therapy with PXD101
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that could compromise compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with PXD101
* HIV-positive patients are ineligible
* Patients with a marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval 500 msec), Long QT Syndrome, or the required use of concomitant medication on PXD101 infusion days that may cause Torsade de Pointes (including disopyramide, dofetilide, ibutilide, procainamide, quinidine, sotalol, bepridil, amiodarone, arsenic trioxide, cisapride, lidoflazine, clarithromycin, erythromycin, halofantrine, pentamidine, sparfloxacin, domperidone, droperidol, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, and methadone)
* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, congestive heart failure related to primary cardiac disease, a condition requiring anti-arrhythmic therapy, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Foon, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

REFERENCES:
- [Derived] Kirschbaum MH, Foon KA, Frankel P, Ruel C, Pulone B, Tuscano JM, Newman EM. A phase 2 study of belinostat (PXD101) in patients with relapsed or refractory acute myeloid leukemia or patients over the age of 60 with newly diagnosed acute myeloid leukemia: a California Cancer Consortium Study. Leuk Lymphoma. 2014 Oct;55(10):2301-4. doi: 10.3109/10428194.2013.877134. Epub 2014 Feb 24. PMID 24369094

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Belinostat)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 78 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Clinical responses were measured according to International Working Group criteria. Bone marrow studies were repeated at a minimum of every three cycles. Per International Working Group criteria: Complete Response (CR): Repeat bone marrow show <5% myeloblasts, and peripheral blood evaluations lasting >=2 months of hemoglobin(>110 g/L), neutrophils(>=1.5x10^9/L), platelets(>=100x10^9/L), blasts (0%) and no dysplasia
Time Frame: Up to 1 year
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 12
percentage of subjects | 0

2. Secondary Outcome: Overall Survival
Description: Survival endpoints will be summarized by the method of Kaplan-Meier
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 12
Months | 9.1 [0.5 to 13.5]

3. Secondary Outcome: Duration of Response
Description: From time of documented treatment response (CR or PR) until progression of death. Complete Response (CR): Repeat bone marrow show <5% myeloblasts, and peripheral blood evaluations lasting >=2 months of hemoglobin(>110 g/L), neutrophils(>=1.5x10^9/L), platelets(>=100x10^9/L), blasts (0%) and no dysplasia. Partial Resonse (PR): requires the same hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to a post-treatment value of 5% to 25% in the bone marrow aspirate. (If the pre-treatment blast percentage was 50-100%, this must decrease to a value between 5-25%. If the pre-treatment blast percentage was 20-49%, this must decrease by at least half to a value greater than 5%.) A value ≤ 5% is also considered a PR if Auer rods are present.
Time Frame: Up to 1 year
Population: There were no formal CRs or PRs seen among the first cohort of 12 patients, resulting in the study's closure. As a result data were not collected.The study was completed as planned and stopped due to futility as written per protocol. It was not terminated prematurely as accrual proceeded per protocol.
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity Summary
Description: Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grade 3 and above toxicities possibly, probably or definitely related to treatment.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 12
participants
  Grade 3 : Dehydration | 1
  Grade 3 : Febrile neutropenia | 1
  Grade 3 : Hematoma | 0
  Grade 3 : Mucositis/stomatitis | 1
  Grade 3 : Nausea | 1
  Grade 3 : Prolonged QTc interval | 1
  Grade 3 : Sodium, serum-low | 1
  Grade 4 : Dehydration | 0
  Grade 4 : Febrile neutropenia | 0
  Grade 4 : Hematoma | 1
  Grade 4 : Mucositis/stomatitis | 0
  Grade 4 : Nausea | 0
  Grade 4 : Prolonged QTc interval | 0
  Grade 4 : Sodium, serum-low | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 12 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Belinostat)
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Belinostat) (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (3)
Electrocardiogram QTc interval prolonged (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Belinostat) (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (27)
Atrial fibrillation (Cardiac disorders) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (15)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 2 (2)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (9)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (15)
Fever (General disorders) | 3 (6)
Flu-like symptoms (General disorders) | 2 (4)
Sinusitis (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 5 (13)
Alkaline phosphatase increased (Investigations) | 3 (14)
Aspartate aminotransferase increased (Investigations) | 4 (14)
Creatinine increased (Investigations) | 4 (9)
Hyperbilirubinemia (Investigations) | 2 (9)
INR increased (Investigations) | 1 (1)
Leukopenia (Investigations) | 2 (6)
Lymphopenia (Investigations) | 4 (9)
Neutrophil count decreased (Investigations) | 6 (22)
Platelet count decreased (Investigations) | 7 (23)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (19)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (7)
Hyponatremia (Metabolism and nutrition disorders) | 5 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (5)
Mental status changes (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (4)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less